CLINICAL TRIAL: NCT06737120
Title: Comparison of Conventional and Modified Free Gingival Graft Techniques in Treating Mandibular Incisor Gingival Recession: a Randomized Clinical Study
Brief Title: Effect of Modified Free Gingival Graft and Conventional Free Gingival Graft on Gingival Recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AYSE HUMEYRA ORUC (Other)
Responsible Party: Sponsor-Investigator, AYSE HUMEYRA ORUC, research assistant, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ModifiedFreeGingivalGraft
Record Dates: First submitted 2024-12-03; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Gingival Recession, Localized; Keratinized Tissue; Free Gingival Graft
Keywords: modified free gingival graft; free gingival graft; gingival recession
MeSH Terms: conditions — Gingival Recession | interventions — fibrinopeptides gamma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- modified free gingival graft (Experimental): A connective tissue pedicle flap will be applied before a free gingival graft is placed in the recipient area.
  Interventions: Procedure: Mod-fgg
- traditional free gingival graft (Experimental)
  Interventions: Procedure: Fgg

INTERVENTIONS:
Procedure: Mod-fgg — Following an intrasulcular incision, 2 mm long horizontal incisions will be made on each side at the level of the gum line. From these incisions, divergent vertical release incisions will be made extending towards the alveolar mucosa. To prepare the recipient area, a thin partial thickness flap will be lifted and then removed. A foil template will be obtained by measuring the dimensions of the resulting area.
  A horizontal incision will be made apical to the exposed root area of the target teeth at a distance corresponding to the height of the exposed root surface. Starting from the endpoints of this incision, two more slightly divergent incisions will be made in the coronal direction. Thus, a connective tissue pedicle flap will be formed and carefully separated from the periosteum. The pedicle graft will be turned over the exposed root surface and fixed with bioabsorbable sutures. The palatal graft will be sutured to cover the connective tissue.
  Arms: modified free gingival graft
Procedure: Fgg — The surgical procedures to be performed in this group will be the same as in the modified free gingival graft group, but no connective tissue pedicle flap will be performed.
  Arms: traditional free gingival graft

SUMMARY:
The aim of this clinical study is to understand whether the modified free gingival graft technique is superior to the conventional free gingival graft:

Will gingival recession completely close in modified free gingival grafting areas? Will there be a significant increase in the amount of keratinized gingiva in modified free gingival grafting participants compared to traditional free gingival grafting participants? Participants will visit our clinic in the 1st, 3rd and 6th months. Necessary clinical parameter measurements will be made by the clinician.

DETAILED DESCRIPTION:
This study will include individuals who come to Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology for various reasons and agree to participate in the study (those who sign the 'informed consent form'). Radiographic and clinical evaluations are routinely performed during the periodontal examination of each patient applying to the periodontology clinic, and routine periodontal status records are taken and archived before and after each planned treatment.

The study was designed as a randomised controlled clinical trial in which 30 patients underwent free gingival grafting (FGG) operation and 30 patients underwent modified free gingival grafting operation (mod-FG). Clinical parameters of the patients were planned to be measured 1 week before, 1 month, 3 months and 6 months after the operation.

The following clinical measurements will be taken by a single investigator at baseline (1 week before surgery) and at 1, 3, 6 and 12 months after surgery:

* Gingival Recession Depth: The distance from the enamel-cementum border to the gingival margin will be measured with an accuracy of 0.1 mm.
* Recession width: The horizontal distance from the widest part of the recession at the enamel-cementum junction to the mesial and distal starting borders, measured with an accuracy of 0.1 mm.
* Keratised Tissue Height: The distance from the gingival margin to the mucogingival junction will be measured with an accuracy of 0.1 mm.
* Papil width: The length of the horizontal line connecting the zenith points of two neighbouring teeth, measured with an accuracy of 0.1 mm.
* Papil height: The length of the vertical distance from the papillary apex to the line passing through the zenith points of the teeth, measured with an accuracy of 0.1 mm.
* Tissue thickness: It will be measured 2 mm apical to the gingival margin in the mid-buccal region under topical anaesthesia with a root canal instrument fitted with a rubber stopper and the distance between the tip of the root canal instrument and the rubber stopper will be measured with a digital caliper.
* Pocket Depth: The distance between the base of the pocket and the free gingival margin will be measured with the help of a periodontal Williams probe at six points for each tooth and the pocket depth will be recorded.

After the initial examination, each person will be given individual oral hygiene instructions and will receive professional dental cleaning, root planing and polishing with a low abrasive polishing paste and a rubber band. Surgical treatment will be planned after adequate personal plaque control has been achieved.

The included participants will be randomly allocated into two groups: conventional free gingival graft (FGG, control) or modified free gingival graft (ModFGG, test). Random allocation will be done in a 1:1 ratio based on a computer-generated number list. Under local anaesthesia, the exposed root surfaces will be cleaned with Gracey curettes and rinsed thoroughly with saline. One of the following two procedures will be performed according to group allocation.

The primary outcome will be the reduction in gingival recession. Sample size calculation will be performed using a 5% significance level and 95% power, assuming that the critical difference in gingival recession reduction between the groups at the end of 12 months is 1.7 mm and the standard deviation is 1.2 mm.

Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS) version 23 (IBM Corp., Armonk, NY). Data will be expressed as mean and standard deviation. Data normality will be assessed using the Kolmogorov-Smirnov test. Differences between parameter means in intra-group comparisons of SDG and modSDG groups will be evaluated using One-way ANOVA (Bonferroni post-hoc) test. Differences between the 2 groups in terms of gingival recession, changes in keratinized tissue height and probing depth, and percentage root coverage will be evaluated by regression analysis using time point and group distribution as main and interaction terms. Results will be expressed as predicted values and 95% confidence intervals. p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:-volunteers aged between 18-65 years.

* To be systemically healthy.
* Not smoking.
* Individuals aged 18 years and over.
* Shallow vestibule (≤5 mm).
* The periodontal pocket depth of the tooth/teeth to be treated should be ≤3 mm and the degree of tooth mobility should be ≤1.
* There should be no cervical composite restoration and no caries-free lesions on the teeth to be treated.
* Presence of Cairo Type 1 class gingival recession on the buccal surface of at most 2 of the mandibular incisors.

Exclusion Criteria:

* pregnancy
* untreated periodontal disease
* parafunctional habits
* poor oral hygiene (persistent whole mouth plaque index > 20%)
* iodine allergy
* excessive dental crowding or misalignment of teeth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
measurement of preoperative periodontal parameters | Preoperatively, before the start of treatment.
  To determine the baseline condition, preoperative measurement of periodontal parameters (amount of keratinized tissue, papilla height, papilla width, probing pocket depth, amount of recession, tissue thickness) will be recorded in millimeters using a periodontal probe.
Preoperative Intraoral Photographs Capture and Evaluation | Preoperatively, before the start of treatment.
  Intraoral photographs of patients will be taken before surgery. These photographs will be used to meet the situation before and after treatment. The photographs will be taken with a high-performance digital camera under standardized angles and lighting.
  Unit of Measurement:
  General condition of oral structures (% change rate).
gingival index measurement | Preoperatively, before the start of treatment.
  The status of gingival health will be assessed using the Gingival Index (Loe and Silness, 1963). This measurement will be made to determine the degree of gingival inflammation and will be scored on a scale from 0 (healthy gingiva) to 3 (severe inflammation and bleeding).
  Unit of Measurement: 0-3 scale.
Plaque Index (PI) measurement | Preoperatively, before the start of treatment.
  The degree of plaque accumulation on the tooth surfaces will be assessed using the Plaque Index (Silness and Loe, 1964). The assessment will be made on a scale from 0 (no plaque) to 3 (entire tooth surface covered with plaque). This measurement will be used to objectively determine the degree of plaque formation.Unit of Measurement: 0-3 scale.

SECONDARY OUTCOMES:
Measurement of Periodontal Parameters | 1,3 and 6 months post-operation.
  Postoperative measurement of periodontal parameters will be recorded using a periodontal probe in millimeters at 1, 3 and 6 months. The parameters include the amount of keratinized tissue, papilla height, papilla width, probing pocket depth , the amount of recession and tissue thickness.
Post-Operative Photographing and Evaluation | 1,3 and 6 months post-operation.
  After surgery, intraoral photographs of patients will be taken at 1, 3 and 6 months. These photographs will be used to analyze the changes that occur after treatment. The photographs will be taken with a high-resolution digital camera under standardized angles and lighting conditions. The evaluation will be performed using specific parameters to measure aesthetic and functional changes.Unit of Measurement:General condition of oral structures (% change rate).
gingival index measurement | 1,3 and 6 months post-operation.
  The status of gingival health will be assessed using the Gingival Index (Loe and Silness, 1963). This measurement will be made to determine the degree of gingival inflammation and will be scored on a scale from 0 (healthy gingiva) to 3 (severe inflammation and bleeding).
  Unit of Measurement: 0-3 scale.
Plaque Index (PI) measurement | 1,3 and 6 months post-operation.
  The degree of plaque accumulation on tooth surfaces will be assessed using the Plaque Index (Silness and Loe, 1964). The measurement will be made on a scale from 0 (no plaque) to 3 (entire tooth surface covered with plaque). This index will be used to evaluate oral hygiene and treatment effectiveness.
  Measurement Unit: 0-3 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camargo PM, Melnick PR, Kenney EB. The use of free gingival grafts for aesthetic purposes. Periodontol 2000. 2001;27:72-96. doi: 10.1034/j.1600-0757.2001.027001072.x. No abstract available. PMID 11551301
- [Background] Carcuac O, Trullenque-Eriksson A, Derks J. Modified free gingival graft technique for treatment of gingival recession defects at mandibular incisors: A randomized clinical trial. J Periodontol. 2023 Jun;94(6):722-730. doi: 10.1002/JPER.22-0581. Epub 2023 Jan 30. PMID 36627509